CLINICAL TRIAL: NCT03700424
Title: The Use of Intravenous Trehalose to Reduce Vascular Inflammation in Acute Coronary Syndrome
Brief Title: Inflammation Reduction by TREhalose AdminisTration
Acronym: IR-TREAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amirhossein Sahebkar, Assistant Professor at Mashhad University of Medical Sciences, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 964334
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Trehalose; Arterial inflammation; Autophagy
MeSH Terms: conditions — Acute Coronary Syndrome; Arteritis | interventions — Trehalose; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be performed double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trehalose (Experimental): Participants will be received intravenous trehalose infusion weekly (15 g/week) for a period of 12 weeks
  Interventions: Drug: Trehalose
- Placebo (Placebo Comparator): Participants will be received equal volume of normal saline weekly for a period of 12 weeks
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Trehalose — Trehalose is a natural disaccharide sugar found extensively among miscellaneous organisms including bacteria, plants, insects, yeast, fungi, and invertebrates. By preventing protein denaturation, it plays various protective roles against stress conditions such as heat, freeze, oxidation, desiccation and dehydration. Owing to this capacity, trehalose is an FDA-approved pharmaceutical excipient that is used as a stabilizer in numerous medicines including parenteral products.
  In this study, all injections will be conducted by a trained nurse in the presence of a specialist physician at a duration of 45-90 minutes.
  Other Names: Mycose
  Arms: Trehalose
Drug: Normal saline — A solution of 0.90% w/v of sodium chloride (NaCl) in water
  Other Names: Physiological saline; Isotonic saline
  Arms: Placebo

SUMMARY:
Arterial wall inflammation has been consistently suggested to serve a causal role in promoting atherosclerosis and predisposing to hard cardiovascular outcomes. Therefore, there is a global trend in the pharmaceutical industry to develop safe and effective anti-inflammatory agents that could lessen arterial wall inflammation and prevent its detrimental impact on atheroma growth and instability. To this end, autophagy has emerged as a key regulator of inflammation and dysfunctional autophagy machinery has been consistently reported as a contributing factor to atherosclerosis and inflammation. Trehalose, a natural disaccharide sugar found extensively among miscellaneous organisms, by preventing protein denaturation plays various protective roles against stress conditions. Numerous studies indicated trehalose's ability to induce macrophage autophagy-lysosomal biogenesis and reduce inflammation. Also, intravenous (IV) administration of trehalose showed beneficial effects in the reversal of atherosclerosis in atherosclerotic animals. Therefore, in this study, the investigators will explore the potential efficacy of IV trehalose administration on arterial inflammation by employing an positron emission tomography (PET) with 18F-labeled fluoro-2-deoxyglucose (18F-FDG) and computed tomography (18F-FDG PET/CT) technique which noninvasively characterizes vascular inflammation and atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18-55 years
* Having a history of acute coronary syndrome
* Having a baseline high-sensitivity C-reactive protein (hs-CRP) of ≥ 2mg/L
* Willingness to participate in the trials.

Exclusion Criteria:

* Lactation or breastfeeding
* Diabetes mellitus
* Nephrotic syndrome or Estimated Glomerular Filtration Rate (eGFR) < 30/mL/min/1.73m2
* Active or recurrent hepatic disease or/and alanine aminotransferase (ALT)/aspartate aminotransferase (AST) (ALT/AST) of > 3 times upper normal limit or total bilirubin of > 2 times upper normal limit
* Active infectious or febrile disease
* Any type of malignancy
* History of transplantation
* Consumption of immunosuppressive drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Arterial wall inflammation in the aorta and carotid arteries | At the beginning and end of the intervention trial (Day 0 and week 12)
  This will be assessed using the 18F-FDG PET/CT imaging technique

SECONDARY OUTCOMES:
Carotid intima-media thickness (cIMT) | At the beginning and end of the intervention trial (Day 0 and week 12)
  This will be assessed using doppler sonography
Measuring beclin-1 to assess autophagy activation | At the beginning and end of the intervention trial (Day 0 and week 12)
Measuring high-sensitivity C-reactive protein (hs-CRP) to assess systemic inflammation | At the beginning and end of the intervention trial (Day 0 and week 12)
Measuring complete blood count (CBC) (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
Assessing lipid profile (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
  Including triglyceride (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C)
Assessing glucose (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
  Fasting blood glucose (FBS)
Measuring thyroid-stimulating hormone (TSH) to assess thyroid function (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
Measuring alanine aminotransferase (ALT), aspartate aminotransferase (AST) and bilirubin (Bil) to assess liver function (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
Measuring creatinine (Cr), urine (Ur) and blood urea nitrogen (BUN) to assess renal function (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
Evaluating electrocardiogram (ECG) and heart rhythm to assess heart function (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)
Measuring creatinine phosphokinase (CPK) to detect muscle damage (Safety) | At the beginning and end of the intervention trial (Day 0 and week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghaem Educational, Research and Treatment Center, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Libby P. Inflammation in atherosclerosis. Arterioscler Thromb Vasc Biol. 2012 Sep;32(9):2045-51. doi: 10.1161/ATVBAHA.108.179705. PMID 22895665
- [Background] Libby P, Hansson GK. Taming Immune and Inflammatory Responses to Treat Atherosclerosis. J Am Coll Cardiol. 2018 Jan 16;71(2):173-176. doi: 10.1016/j.jacc.2017.10.081. No abstract available. PMID 29325641
- [Background] Liao X, Sluimer JC, Wang Y, Subramanian M, Brown K, Pattison JS, Robbins J, Martinez J, Tabas I. Macrophage autophagy plays a protective role in advanced atherosclerosis. Cell Metab. 2012 Apr 4;15(4):545-53. doi: 10.1016/j.cmet.2012.01.022. Epub 2012 Mar 22. PMID 22445600
- [Background] Maiuri MC, Grassia G, Platt AM, Carnuccio R, Ialenti A, Maffia P. Macrophage autophagy in atherosclerosis. Mediators Inflamm. 2013;2013:584715. doi: 10.1155/2013/584715. Epub 2013 Jan 21. PMID 23401644
- [Background] Shao BZ, Han BZ, Zeng YX, Su DF, Liu C. The roles of macrophage autophagy in atherosclerosis. Acta Pharmacol Sin. 2016 Feb;37(2):150-6. doi: 10.1038/aps.2015.87. Epub 2016 Jan 11. PMID 26750103
- [Background] Iwatsuka R, Matsue Y, Yonetsu T, O'uchi T, Matsumura A, Hashimoto Y, Hirao K. Arterial inflammation measured by 18F-FDG-PET-CT to predict coronary events in older subjects. Atherosclerosis. 2018 Jan;268:49-54. doi: 10.1016/j.atherosclerosis.2017.11.016. Epub 2017 Nov 21. PMID 29175654
- [Background] Chrapko BE, Chrapko M, Nocun A, Stefaniak B, Zubilewicz T, Drop A. Role of 18F-FDG PET/CT in the diagnosis of inflammatory and infectious vascular disease. Nucl Med Rev Cent East Eur. 2016;19(1):28-36. doi: 10.5603/NMR.2016.0006. PMID 26841377
- [Background] Menezes LJ, Kotze CW, Hutton BF, Endozo R, Dickson JC, Cullum I, Yusuf SW, Ell PJ, Groves AM. Vascular inflammation imaging with 18F-FDG PET/CT: when to image? J Nucl Med. 2009 Jun;50(6):854-7. doi: 10.2967/jnumed.108.061432. Epub 2009 May 14. PMID 19443587
- [Background] Chen Q, Haddad GG. Role of trehalose phosphate synthase and trehalose during hypoxia: from flies to mammals. J Exp Biol. 2004 Aug;207(Pt 18):3125-9. doi: 10.1242/jeb.01133. PMID 15299033
- [Background] Castillo K, Nassif M, Valenzuela V, Rojas F, Matus S, Mercado G, Court FA, van Zundert B, Hetz C. Trehalose delays the progression of amyotrophic lateral sclerosis by enhancing autophagy in motoneurons. Autophagy. 2013 Sep;9(9):1308-20. doi: 10.4161/auto.25188. Epub 2013 Jun 6. PMID 23851366
- [Background] Mardones P, Rubinsztein DC, Hetz C. Mystery solved: Trehalose kickstarts autophagy by blocking glucose transport. Sci Signal. 2016 Feb 23;9(416):fs2. doi: 10.1126/scisignal.aaf1937. PMID 26905424
- [Background] Sergin I, Evans TD, Zhang X, Bhattacharya S, Stokes CJ, Song E, Ali S, Dehestani B, Holloway KB, Micevych PS, Javaheri A, Crowley JR, Ballabio A, Schilling JD, Epelman S, Weihl CC, Diwan A, Fan D, Zayed MA, Razani B. Exploiting macrophage autophagy-lysosomal biogenesis as a therapy for atherosclerosis. Nat Commun. 2017 Jun 7;8:15750. doi: 10.1038/ncomms15750. PMID 28589926
- [Background] van der Valk FM, Bekkering S, Kroon J, Yeang C, Van den Bossche J, van Buul JD, Ravandi A, Nederveen AJ, Verberne HJ, Scipione C, Nieuwdorp M, Joosten LA, Netea MG, Koschinsky ML, Witztum JL, Tsimikas S, Riksen NP, Stroes ES. Oxidized Phospholipids on Lipoprotein(a) Elicit Arterial Wall Inflammation and an Inflammatory Monocyte Response in Humans. Circulation. 2016 Aug 23;134(8):611-24. doi: 10.1161/CIRCULATIONAHA.116.020838. Epub 2016 Aug 5. PMID 27496857
- [Background] van der Valk FM, Verweij SL, Zwinderman KA, Strang AC, Kaiser Y, Marquering HA, Nederveen AJ, Stroes ES, Verberne HJ, Rudd JH. Thresholds for Arterial Wall Inflammation Quantified by 18F-FDG PET Imaging: Implications for Vascular Interventional Studies. JACC Cardiovasc Imaging. 2016 Oct;9(10):1198-1207. doi: 10.1016/j.jcmg.2016.04.007. Epub 2016 Sep 14. PMID 27639759